CLINICAL TRIAL: NCT04845867
Title: Thyroid HEmorrhage DetectOr Study
Brief Title: A Prospective, Single-arm, Multi-centre, Blinded, Observational, Diagnostic Accuracy Study With a Diagnostic Medical Product
Acronym: HEDOS
Status: Recruiting | Type: Observational
Sponsor: ISAR-M GmbH (Industry)
Collaborators: CRI-The Clinical Research Institute GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: HEDOS-2021
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Thyroid
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Measurement and digital documentation: continuous measurement and digital documentation with alarms and display off
  Interventions: Device: ISAR-M THYRO

INTERVENTIONS:
Device: ISAR-M THYRO — A diagnostic device for early detection of haemorrhage following thyroid surgery

SUMMARY:
After thyroid surgery, 0.6 to 4% of patients develop postoperative bleeding. 90% of this postoperative bleeding occurs within the first 48 hours. Most of the time, the complications are rapidly progressing and require immediate attention. Up to 0.6% of patients with postoperative bleeding die. In a clinical study with postoperative pressure measurements it could be shown that postoperative bleeding without interruption leads to a continuous increase in pressure in the neck, as is observed when coughing and pressing. Systematic invasive pressure measurement in the thyroid compartment after surgery might detect a continuous increase in pressure which is often caused by a growing haematoma, indicating serious post-surgery bleeding at a much earlier time compared to state of the art diagnostic workflow. n routine clinical care, detection of serious haemorrhage depends on the patients alerting symptoms even if post-operative intermittent monitoring of vital parameters and wound conditions is performed according to current medical guidelines and local instructions. Device-based, continuous haemorrhage detection within 36 to 48 hours after surgery would allow to objectively measure an increase in cervical pressure before symptoms occur, i.e. early detection of risk leading to timely therapeutic actions. Thus, the risk of serious complications like hypoxic brain damage and death caused by post-operative haemorrhage is minimized. In addition, the intervention team would be able to fine-tune necessary actions during the rescue procedure based on objective pressure values, e.g. the decision to open cutaneous sutures immediately or later in the operation theatre, and therefore reduce additional perioperative morbidity and increase patients' safety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Indication for thyroid surgery (e.g. total thyroidectomy, subtotal resection, partial resection or lobectomy) in routine clinical care according to applicable medical guidelines using all adequate surgical approaches.
* Signed informed consent

Exclusion Criteria:

- Intended use of drains

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HEDOS will enrol and measure presumably 1,470 eligible adult patients and follow each of them for 1 month, assuming that 22 cases of clinically relevant haemorrhage within 48 hours following thyroid surgery will be observed. It will be conducted in Germany and Austria with about 50 clinical sites participating.
Sampling Method: Non-Probability Sample
Enrollment: 1470 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-10-23 (Estimated); Study Completion 2024-11-24 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity | within 48 hours following thyroid surgery
  detection of clinically relevant haemorrhage compared to the gold standard of detection in routine clinical care using 15 mmHg as cut-off
Sensitivity and specificity | within 48 hours following thyroid surgery
  Sensitivity and specificity of detection of clinically relevant haemorrhage within 48 hours following thyroid surgery compared to the gold standard of routine clinical care detection in a three-level decision system using 10 and 20 mmHg as cut-offs

SECONDARY OUTCOMES:
Specificity | within 48 hours following thyroid surgery
  Specificity as well as positive and negative predictive values of detection of clinically relevant haemorrhage within 48 hours following thyroid surgery compared to the gold standard of detection in routine clinical care using the two-level and the three-level decision system.following thyroid surgery compared to the gold standard of routine clinical care detection in routine clinical care using the two-level and three-level decision system
Safety of the use of ISAR-M THYRO | 1 month
  Safety of the use of ISAR-M THYRO by means of adverse events within 1 month following thyroid surgery

CONTACTS AND LOCATIONS:
Overall Officials: Markus MA Albertsmeier, Dr., Study Chair — Clinic for General, Visceral, Vascular and Transplant Surgery - Großhadern Campus,
Locations (1):
- Krankenhaus Agatharied, Hausham, Germany

IPD SHARING:
Plan to Share IPD: Undecided